CLINICAL TRIAL: NCT05045989
Title: Mixed-methods Process Evaluation of a Residence-Based SARS-CoV-2 Testing Participation Pilot on a UK University Campus During the COVID-19 Pandemic.
Brief Title: Process Evaluation of a Residence-Based SARS-CoV-2 Testing Participation Pilot
Acronym: RB-TPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Holly Blake, Associate Professor of Behavioural Sciences, University of Nottingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FMHS 96-0920
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Testing

STUDY DESIGN:
Intervention Model Description: Process evaluation of a SARS-CoV-2 testing participation uptake scheme in a single group of students living in two halls of residence.
Masking Description: N/A process evaluation, single group intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Residence-based asymptomatic SARS-CoV-2 testing (Experimental): The aim of the RB-TPP was to increase and maintain participation of students in regular COVID-19 testing in university residences. The R-TPP was delivered over 4 weeks in April-May 2021 and required asymptomatic students to take a saliva test for COVID-19, twice weekly for four weeks. This was combined with relaxed social restrictions within the residence during the study period (i.e., removing the need for 2 metre distancing between students living in the same residence), surge testing and enhanced support for students who were required to self-isolate (i.e., welfare and financial support).
  Interventions: Behavioral: Residence-based testing participation pilot (SARS-CoV-2 testing with relaxed social distancing restrictions)

INTERVENTIONS:
Behavioral: Residence-based testing participation pilot (SARS-CoV-2 testing with relaxed social distancing restrictions) — SARS-CoV-2 asymptomatic saliva testing (as available to all students at staff at the participating university) delivered with relaxed social distancing (behavioural element) in two halls of residence.

SUMMARY:
Mixed-methods process evaluation of a residence-based asymptomatic SARS-CoV-2 testing participation pilot

DETAILED DESCRIPTION:
Regular testing for SARS Coronavirus 2 (SARS-CoV-2) is an important strategy for controlling virus outbreaks on university campuses during the COVID-19 pandemic but testing participation rates can be low. The Residence-Based Testing Participation Pilot (RB-TPP) was a novel intervention implemented at two student residences on a large university campus in the UK over four weeks. The aim of the pilot was to increase the frequency of asymptomatic SARS-CoV-2 saliva testing onsite. This process evaluation aimed to determine whether RB-TPP was implemented as planned and identify implementation barriers and facilitators. A mixed-methods process evaluation was conducted alongside the RB-TPP. Evaluation participants were students (who opted in, or out of the RB-TPP) and staff with a role in service provision or student support. Monitoring data were collected from the intervention delivery team and meeting records. Data were collected from students via an online survey (n=152) and seven focus groups (n=30), and from staff via individual interviews (n=13). Quantitative data were analysed descriptively and qualitative data thematically.

ELIGIBILITY:
Inclusion Criteria:

* Student is living in one of the two participating halls of residence.
* staff with operational or student support role.
* consents to participate.

Exclusion Criteria:

* Student is not living in the hall of residence at the start of the RB-TPP.
* does not consent to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Reach | 1 week
  Program reach was evaluated through the number of students recruited into the RB-TPP compared to the number of potentially eligible students living in one of the two participating sites in April 2021

SECONDARY OUTCOMES:
Adherence | 4 weeks
  Participant adherence was defined as the proportion of students who completed all tests offered.
Dose | 4 weeks
  Number of tests offered
Generalised Anxiety Disorders Scale (Spitzer et al., 2006; Kroenke et al., 2007). | 4 weeks
  A 7-item anxiety scale with good reliability, as well as criterion, construct, factorial, and procedural validity. A cut point of >=10 indicates moderate to severe anxiety. Higher scores indicate higher anxiety.
Student Focus Groups | 4 weeks
  Student's views towards the RB-TPP. Small group discussions lasting approximately 60 mins conducted at mid-point and/or programme end.
Staff interviews | 4 weeks
  Staff views towards the RB-TPP. Individual interviews lasting approximately 20-60 mins conducted at programme end.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Blake, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analysed during the current study are not publicly available due to risk of identification of participants and service providers but are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Blake H, Somerset S, Mahmood I, Mahmood N, Corner J, Ball JK, Denning C. A Qualitative Evaluation of the Barriers and Enablers for Implementation of an Asymptomatic SARS-CoV-2 Testing Service at the University of Nottingham: A Multi-Site Higher Education Setting in England. Int J Environ Res Public Health. 2022 Oct 12;19(20):13140. doi: 10.3390/ijerph192013140. PMID 36293719
- [Derived] Blake H, Carlisle S, Fothergill L, Hassard J, Favier A, Corner J, Ball JK, Denning C. Mixed-methods process evaluation of a residence-based SARS-CoV-2 testing participation pilot on a UK university campus during the COVID-19 pandemic. BMC Public Health. 2022 Aug 2;22(1):1470. doi: 10.1186/s12889-022-13792-8. PMID 35915479